CLINICAL TRIAL: NCT06275984
Title: Effectiveness of Online Training in Cardiopulmonary Resuscitation Maneuvers for a Network of Volunteers to Increase Survival in Cardiac Arrest. EFORCP Study
Brief Title: Effectiveness of Online Training in Cardiopulmonary Resuscitation Maneuvers for a Network of Volunteers.
Acronym: EFORCP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PI23/00288; 4R23/440 (Other: IDIAP Jordi Gol)
Record Dates: First submitted 2024-02-09; First posted 2024-02-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Cardiorespiratory Arrest; Cardiopulmonary Arrest With Successful Resuscitation
Keywords: Heart Arrest; Simulation Training; Primary Health Care; Defibrillators
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Online training (Other): Participants will perform an online training in CPR-AED
  Interventions: Other: online CPR-AED training

INTERVENTIONS:
Other: online CPR-AED training — The online CPR-AED training consists of successfully completing the online training course. To access the course, interested persons must register on a Moodle environment platform, with free and open access, through the following link: https://register.magnore.com/registre-curs-de-reanimacio -cardiopulmonary-dea/
  Online training takes 3-4h and the participant will have access for 1 month (7x24h).

SUMMARY:
Background: Cardiorespiratory arrest (CPA) occurs when there is a cessation of cardiac mechanical activity, typically diagnosed by the absence of consciousness, pulse, and breathing. Actions taken in response to CPA include recognizing the condition and promptly notifying emergency medical services, initiating Cardiopulmonary Resuscitation (CPR) maneuvers, and employing an Automated External Defibrillator (AED). Survival rates are directly influenced by the time elapsed between CPA onset and the initiation of CPR maneuvers, as well as the quality of these interventions

Hypotheses: Online education in CPR maneuvers is an effective and efficient tool for training individuals from the general population on how to respond to cardiac arrests

Objectives: The primary aim of this study is to assess the efficacy of online CPR and AED training within the general population of the province of Tarragona. Specific objectives include: 1) evaluating participants' theoretical and practical CPR skills in the short and medium term following online training, and 2) exploring the experiences of individuals who have completed the online training and simulation sessions using qualitative methodology.

Methodology:This study will unfold in several phases: 1) Online CPR-AED training and assessment of theoretical knowledge acquisition; 2) Evaluation of acquired practical CPR skills (know-how) within a simulation environment, conducted on a subset of the population completing phase 1;3)Analysis of the experiences of a subset of individuals who have participated in the preceding two phases, employing qualitative methodology

Variables and determinations:The primary response variable for phase 1 will be the difference in scores obtained from the online questionnaire between the final (post-training) and initial (pre-training) assessments.

In phase 2, the main variable will be the pass/fail categorization of scores in the simulation. This evaluation will be conducted by two members of the Advanced Clinical Simulation Unit at Joan XXII Hospital using a predefined checklist. Throughout the various phases of the study, socio-demographic data and course performance data will be taken into account

Expected results: The research team for this study aims to ascertain the efficacy and effectiveness of online CPR-AED training within the general population. Furthermore, the study aims to provide evidence regarding the optimal duration and frequency for repeating such training.

Applicability and Relevance: This proposal advocates for a significant and innovative project, given the dearth of literature on this topic. While there are existing indications and studies on CPR-AED training among specific populations such as students and healthcare professionals, the presented proposal seeks to broaden the scope of training to encompass the general population.

DETAILED DESCRIPTION:
Study Development:

The recruitment period spans from June 2024 to June 2025. Individuals meeting the selection criteria will have access to the online training. Upon registration, they will be notified of the study's existence, and if they consent, their data may be analyzed in phase 1. Participants will also be informed about phase 2 and asked for their interest in participating. Those interested will need to provide contact information (telephone and/or email).

For phase 2, a random sample will be drawn from individuals expressing interest in the simulation. All participants in this phase will receive an information sheet and will be required to sign an informed consent form.

Phase 1: Online CPR and AED Training and Evaluation of Theoretical Skills

Participants will be administered a questionnaire on CPR-AED knowledge before and after completing the online training. This questionnaire, tailored specifically for the course, adheres to the recommendations of the Spanish Cardiopulmonary Resuscitation Council. It comprises five questions in various formats (e.g., multiple-choice, sequencing actions). To obtain the training certificate, participants must answer all five questions correctly, with unlimited attempts permitted. The primary response variable for this phase will be the difference between the final score (on the first attempt) and the initial score. Additionally, the number of attempts made until achieving the maximum score (5) will be recorded as a variable

Phase 2: Evaluation of Practical Skills Acquired afetr the online training through Simulations

Monthly evaluations will be conducted at the Advanced Clinical Simulation Unit of HJ23 (Hospital Universitari Joan XXIII), with 15 participants per session. This structure ensures that three random samples of 52 individuals each will be evaluated at 3, 6, and 12 months following completion of the online training.

To assess phase 2 (simulation), two evaluators from the Advanced Clinical Simulation Unit of HJ23, who are independent of the research team, will complete a checklist based on their observations of the participants' performance during the evaluation. The evaluation will be considered successful if the participant adequately performs eight out of nine actions on the checklist, with a high agreement between evaluators (Kappa index greater than 0.8). The primary response variable for this practical assessment will be the percentage of participants who pass the test. Additionally, the time elapsed between completion of the online training and the simulation will be recorded.

Statistical Analysis:

A descriptive analysis of the study population will be conducted for both participants in phase one and the subsample undertaking simulations. Continuous variables will be presented as mean (± standard deviation) or median and interquartile range (IQR), while categorical variables will be expressed as absolute and relative frequencies.

To compare scores in the pre- and post-training tests (phase 1), the Student's t-test for related samples or the non-parametric Wilcoxon test will be utilized.

For phase 2, absolute and relative frequencies of individuals passing tests (overall and by period) will be provided, along with 95% confidence intervals. Additionally, the success percentage for each assessed item will be analyzed. These scores will be compared across different periods (3, 6, and 12 months) using the Chi-square or Fisher's exact test if necessary.

Furthermore, multivariate regression models will be explored, with the response variable being the dichotomous pass/fail variable (binary logistic regression) in phase 2, and including other study variables as adjustment variables. Crude and adjusted odds ratios (ORs) will be provided for all variables included in the final models. This analysis aims to identify variables associated with succes obtained in the simulation (phase 2).

The threshold for statistical significance is set at p<0.05. All statistical analyses will be performed using the R Statistics program (R Foundation for Statistical Computing, Vienna, Austria; version 4.1.2 or later).

Phase 3: Evaluation of Participants' Experience

For the qualitative study, interviews will be conducted with focus groups consisting of four to six individuals, selected based on representativeness criteria, from those who have completed both previous phases (online training and simulation). The objective of this phase is to gain insight into participants' experiences and, based on these insights, to adapt and enhance the online training program. Participants will be asked about the strengths and weaknesses of the training and assessments in both phases, and will be encouraged to provide suggestions for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Residents in the municipalities of Camp de Tarragona
* With internet access

Exclusion Criteria:

* Language difficulties
* Disability that prevents the correct completion or performance of a CPR maneuver (exclusion criteria for moving to phase 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Difference between pre and post training scores in ad hoc designed scale | 12 months
  The scale used to measure the acquisition of knowledge through online theoretical training has been designed ad hoc for the present study, following the recommendations of the Spanish Council of Cardiopulmonary Resuscitation. It consists of 5 items. The scoring ranges from 0 to 5, with higher scores indicating greater knowledge.
Percentage of participants that reach or exceed 10 out of 12 on the checklist | 14 months
  Percentage of participants that pass the CPR-AED evaluation in a simulated environment. (phase 2)

SECONDARY OUTCOMES:
Odds ratios (with 95% CI) for adjustment variables | 24 months
  These odds ratios will assess the association between sociodemographic and other study variables and the likelihood of success in the simulation (indicating competence in CPR).
Scores on the standard satisfaction questionnaire commonly used by the Catalan Health Institute to evaluate training activities | 12 months
  The questionnaire used to measure satisfaction is a standard questionnaire commonly employed by the Catalan Health Institute to evaluate the satisfaction of students participating in training activities. It assesses organizational aspects, methodology, applicability, overall assessment (expectations and whether the course is recommendable to others), and the instructors. Each item is rated from 1 to 5. The scoring ranges from 6 to 30. Higher scores indicate a higher degree of satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No